CLINICAL TRIAL: NCT01375036
Title: A Prospective, 5-year Registry Study to Monitor the Susceptibility to Aztreonam of Pseudomonas Aeruginosa (PA) Isolates From Patients With Cystic Fibrosis in the United States [AIR-CF5]
Brief Title: Registry to Monitor the Susceptibility to Aztreonam of Pseudomonas Aeruginosa Isolates From Cystic Fibrosis Patients
Acronym: AIR-CF5
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: GX-US-205-0128
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; PA; Pseudomonas aeruginosa; CF; aztreonam
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pseudomonas aeruginosa isolates from sputum or throat swab specimens
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, longitudinal, 5-year study that will enroll participants from the existing Cystic Fibrosis Foundation (CFF) patient registry. Each enrolled participant will provide samples for microbiological evaluation, obtained upon enrollment and then once per year thereafter for 5 years.

ELIGIBILITY:
Key Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study.

* Current participant or willingness to participate in the CFF patient registry database
* ≥ 6 years of age
* Subject has CF as diagnosed by one of the following

  * Documented sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis test, or
  * Two well-characterized genetic mutations in the CFTR gene, or
  * Abnormal nasal potential difference (NPD) AND accompanying clinical characteristics consistent with CF. For subjects who lack documentation of either a positive sweat chloride test or an abnormal NPD, and who have only one well-characterized genetic mutation of the CFTR gene, the diagnosis of CF is determined by the Investigator.
* FEV1 ≥ 25% predicted and ≤ 90% predicted.
* ≥ 2 lower respiratory tract cultures positive for PA with results documented in the subject's medical history.
* Subject must be able to provide written informed consent/assent prior to any study related procedure; parent/guardian must be able to give written informed consent as necessary prior to any study related procedure.

Key Exclusion Criteria:

Subjects who meet the following exclusion criterion are not to be enrolled in this study.

• Any serious active medical or psychiatric illness that, in the opinion of the Investigator, would interfere with subject assessment.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A representative cross-section of individuals with mild (FEV1 75% to ≤ 90% predicted), moderate (FEV1 40% to 74% predicted), or severe (FEV1 <40% predicted) lung disease and a history of ≥ 2 lower respiratory tract cultures positive for PA (at any time) will be enrolled. This will include approximately 100 individuals with pre-study exposure to Cayston (defined as having received at least one prior 28-day course of Cayston at any time before enrolling into the study). Enrollment will be monitored and potentially modified to ensure that adequate numbers of participants in each disease severity category are included. At the Investigator's discretion, participants enrolled in this study can be allowed to participate in clinical trials with other investigational therapies as appropriate.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2011-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants whose least susceptible Pseudomonas aeruginosa (PA) isolate has a ≥ 4-fold increase in aztreonam minimum inhibitory concentration over 1 year and is above the parenteral breakpoint (> 8 μg/mL) | Up to 5 years
  This proportion will be compared annually over 5 years.

SECONDARY OUTCOMES:
Annual mean change and mean change from baseline in FEV1 (liters) and FEV1 % predicted | Baseline to Year 5
Annual number of hospitalizations and the total number of hospitalizations at the end of each year | Up to 5 years
Annual number of days hospitalized and the total number of hospitalization days at the end of each year | Up to 5 years
Annual mean change and mean change from baseline in body mass index (BMI) | Baseline to Year 5
Annual number of Cayston treatment courses per participant and the total number of Cayston treatment courses at the end of each year in participants that used Cayston | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (30):
- United States (30):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - University of Arizona, Tucson, Arizona
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - The Children's Hospital, Denver, Colorado
  - National Jewish Health, Denver, Colorado
  - Central Florida Pulmonary Group, Altamonte, Florida
  - Nemours Children's Clinic, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospitals & Clinics of Minnesota, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Lung Specialists, Las Vegas, Nevada
  - Albany Medical College, Albany, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinati Children's Hosptial Medical Center, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Keating CL, Zuckerman JB, Singh PK, McKevitt M, Gurtovaya O, Bresnik M, Marshall BC, Saiman L. Pseudomonas aeruginosa Susceptibility Patterns and Associated Clinical Outcomes in People with Cystic Fibrosis following Approval of Aztreonam Lysine for Inhalation. Antimicrob Agents Chemother. 2021 Feb 17;65(3):e02327-20. doi: 10.1128/AAC.02327-20. Print 2021 Feb 17. PMID 33318007